CLINICAL TRIAL: NCT01917006
Title: An Exploratory Study of the Safety and Efficacy of BOTOX® for the Treatment of Premature Ejaculation
Brief Title: A Safety and Efficacy Study of OnabotulinumtoxinA in Premature Ejaculation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic business decision was made to terminate the program. There were no safety concerns.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-133; 2013-001650-94 (EudraCT Number)
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- OnabotulinumtoxinA Dose 1 (Experimental): OnabotulinumtoxinA Dose 1 injected into specified muscle per protocol on Day 1.
  Interventions: Drug: OnabotulinumtoxinA
- OnabotulinumtoxinA Dose 2 (Experimental): OnabotulinumtoxinA Dose 2 injected into specified muscle per protocol on Day 1. Participants were eligible for another treatment after 12 weeks.
  Interventions: Drug: OnabotulinumtoxinA
- OnabotulinumtoxinA Dose 3 (Experimental): OnabotulinumtoxinA Dose 3 injected into specified muscle per protocol on Day 1.
  Interventions: Drug: OnabotulinumtoxinA
- OnabotulinumtoxinA Dose 4 (Experimental): OnabotulinumtoxinA Dose 4 injected into specified muscle per protocol on Day 1.
  Interventions: Drug: OnabotulinumtoxinA
- OnabotulinumtoxinA Dose 5 (Experimental): OnabotulinumtoxinA Dose 5 injected into specified muscle per protocol on Day 1.
  Interventions: Drug: OnabotulinumtoxinA
- OnabotulinumtoxinA Dose 6 (Experimental): OnabotulinumtoxinA Dose 6 injected into specified muscle per protocol on Day 1.
  Interventions: Drug: OnabotulinumtoxinA
- Placebo (Placebo Comparator): Placebo (normal saline) injected into specified muscle per protocol on Day 1.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: OnabotulinumtoxinA — OnabotulinumtoxinA injected into specified muscle per protocol on Day 1.
  Other Names: BOTOX®; Botulinum Toxin Type A
  Arms: OnabotulinumtoxinA Dose 1; OnabotulinumtoxinA Dose 2; OnabotulinumtoxinA Dose 3; OnabotulinumtoxinA Dose 4; OnabotulinumtoxinA Dose 5; OnabotulinumtoxinA Dose 6
Drug: Normal Saline — Placebo (normal saline) injected into specified muscle per protocol on Day 1.
  Arms: Placebo

SUMMARY:
This is a safety and efficacy study of OnabotulinumtoxinA for the treatment of premature ejaculation (PE) in male participants.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, randomized, double-blind, placebo-controlled, dose-escalation study to assess a range of doses of OnabotulinumtoxinA for the treatment of male participants with PE. Participants will attend a minimum of 6 or 7 clinic visits and also have 1 or 2 telephone visits. Partners will need to attend a clinic visit during the screening period to provide informed consent and to receive training on measurement and recording of the intravaginal ejaculatory latency time (IELT). Participants will be enrolled in cohorts. Within the first 5 cohorts, 8 participants are to receive OnabotulinumtoxinA and 2 participants to receive placebo. For cohort 6, 12 participants will receive OnabotulinumtoxinA and 12 participants will receive placebo. Participants will receive a single treatment of study medication delivered bilaterally to the bulbospongiosus muscle. The initial OnabotulinumtoxinA total dose in this dose escalation study will be 5 U and the maximum OnabotulinumtoxinA total dose will be 100 U. Upon request and if eligible, participants in cohort 6, will have the option to receive a second injection of OnabotulinumtoxinA (Open-label).

ELIGIBILITY:
Inclusion Criteria:

* History of premature ejaculation
* Stable monogamous sexual relationship with female partner for at least 6 months, and intends to continue with the same partner for the duration of the study
* Participant has ability to follow study instructions and complete study assessment tools

Exclusion Criteria:

* Premature ejaculation caused by medical or surgical issues, or is related to stress or other issues (eg, relationship problems)
* Pain with ejaculation
* Planned use of topical penile treatments (eg, anesthetics, herbal treatments) or penile injections during the study
* Prior genital, prostatic or lower urinary tract surgery (other than vasectomy or circumcision)
* Previous or current usage of botulinum toxin therapy of any serotype for any urological condition
* Use of botulinum toxin therapy of any serotype for any nonurological condition (eg, cosmetic, chronic migraine) during the 12 weeks prior to screening, or planned usage during the study
* Diagnosis of Myasthenia gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2013-08-07 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Radecki, Study Director — Allergan
Locations (10):
- United States (6):
  - San Diego Sexual Medicine, San Diego, California
  - LA Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Connecticut Clinical Research Center, Middlebury, Connecticut
  - Center for Marital and Sexual Health of South Florida, West Palm Beach, Florida
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Manhattan Medical Research, New York, New York
- United Kingdom (4):
  - Celerion, Belfast
  - King's College Hospital, London
  - Queen Anne Street Medical Center, London
  - St Mary's Hospital, London

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received a single treatment of either placebo or OnabotulinumtoxinA (Doses 1, 2, 3, 4, 5, 6), delivered bilaterally to the bulbospongiosus muscle in randomized-treatment period. Participants who completed 12 weeks of randomized period were eligible to receive second injection with OnabotulinumtoxinA Dose 2 in Open-label Period.
Groups:
- OnabotulinumtoxinA Dose 2 (Open-label Period): Participants who completed 12 weeks of randomized period were eligible to receive a second injection with active drug in the Open-label Period.
Period: Randomized-treatment Period
Arm/Group | OnabotulinumtoxinA Dose 1 | OnabotulinumtoxinA Dose 2 | OnabotulinumtoxinA Dose 3 | OnabotulinumtoxinA Dose 4 | OnabotulinumtoxinA Dose 5 | OnabotulinumtoxinA Dose 6 | Placebo | OnabotulinumtoxinA Dose 2 (Open-label Period)
Started | 5 | 7 | 8 | 8 | 8 | 8 | 15 | 0
Completed | 3 | 7 | 8 | 7 | 8 | 7 | 14 | 0
Not Completed | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Personal Reasons | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Miscellaneous Reasons | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Open-label Period
Arm/Group | OnabotulinumtoxinA Dose 1 | OnabotulinumtoxinA Dose 2 | OnabotulinumtoxinA Dose 3 | OnabotulinumtoxinA Dose 4 | OnabotulinumtoxinA Dose 5 | OnabotulinumtoxinA Dose 6 | Placebo | OnabotulinumtoxinA Dose 2 (Open-label Period)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population included all randomized participants who received study treatment and had post-baseline intravaginal ejaculatory latency time (IELT) data available based on the dose actually received by the participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA Dose 1 | OnabotulinumtoxinA Dose 2 | OnabotulinumtoxinA Dose 3 | OnabotulinumtoxinA Dose 4 | OnabotulinumtoxinA Dose 5 | OnabotulinumtoxinA Dose 6 | Placebo | Total
Number analyzed (Participants) | 5 | 7 | 8 | 7 | 8 | 7 | 15 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (10.83) | 41.9 (11.65) | 39.1 (5.62) | 39.3 (9.05) | 40.1 (6.53) | 39.9 (5.96) | 41.0 (6.08) | 40.4 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 7 | 8 | 7 | 8 | 7 | 15 | 57
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 3 | 4 | 5 | 5 | 5 | 6 | 9 | 37
  Black | 1 | 2 | 1 | 1 | 1 | 0 | 3 | 9
  Asian | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 4
  Hispanic | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 5
  Other | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Geometric Mean Intravaginal Ejaculatory Latency Time (IELT)
Description: IELT, the time from vaginal penetration to ejaculation, was measured by a stopwatch and was recorded in the sexual intercourse diary (SID). The Logarithm Value of the Geometric Mean of each individual participant's IELT recorded in the SID up to each time point was calculated. The mean and standard deviation (SD) of log-transformed geometric mean IELTs are then calculated for each treatment group. An Analysis of Covariance (ANCOVA) Model with treatment as the fixed effect and baseline geometric mean IELT as the covariate was used for analyses. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: The modified intent-to-treat (mITT) population included all randomized participants who received study treatment and had post-baseline intravaginal ejaculatory latency time (IELT) data available based on the dose actually received by the participant. Number analyzed is the number of participants with available data at the given time-point.
Measure: Mean (Standard Deviation); unit: log(seconds)
Arm/Group | OnabotulinumtoxinA Dose 1 | OnabotulinumtoxinA Dose 2 | OnabotulinumtoxinA Dose 3 | OnabotulinumtoxinA Dose 4 | OnabotulinumtoxinA Dose 5 | OnabotulinumtoxinA Dose 6 | Placebo
Number analyzed (Participants) | 5 | 7 | 8 | 7 | 8 | 7 | 15
log(seconds)
  Baseline: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 15
  Baseline | 3.57 (0.283) | 3.50 (0.631) | 3.46 (0.371) | 3.52 (0.531) | 3.53 (0.475) | 3.54 (0.505) | 3.46 (0.610)
  Change from Baseline to Week 12: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 15
  Change from Baseline to Week 12 | 0.55 (1.037) | 0.69 (1.426) | 0.05 (0.856) | 0.30 (0.472) | 0.31 (0.525) | 0.59 (0.719) | 0.44 (0.615)
Statistical Analysis 1: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; Test type: Superiority; p = 0.393, ANCOVA — Least square mean and one-sided p-value of mean difference vs placebo for each active OnabotulinumtoxinA dose level is calculated from analysis of covariance (ANCOVA) Model with treatment as fixed effect and baseline geometric mean IELT as covariate; Least square mean difference = 0.11
Statistical Analysis 2: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; Test type: Superiority; p = 0.263, ANCOVA — Least square mean and one-sided p-value of mean difference vs placebo for each active OnabotulinumtoxinA dose level is calculated from the ANCOVA Model with treatment as the fixed effect and baseline geometric mean IELT as the covariate; Least Square Mean Difference = 0.25
Statistical Analysis 3: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; Test type: Superiority; p = 0.861, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.39
Statistical Analysis 4: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; Test type: Superiority; p = 0.647, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.14
Statistical Analysis 5: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; Test type: Superiority; p = 0.645, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.13
Statistical Analysis 6: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; Test type: Superiority; p = 0.343, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.15

2. Secondary Outcome: Change From Baseline in Average IELT
Description: IELT, the time from vaginal penetration to ejaculation, was measured by a stopwatch and was recorded in the SID. The average of each individual participant's IELT recorded in the SID up to each time point was calculated. The mean and SD of average IELTs were then calculated for each treatment group. An ANCOVA Model with treatment as the fixed effect and baseline average mean IELT as the covariate was used for analyses. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Weeks 2, 4, 6, 8, 10, and 12
Population: The mITT population included all randomized participants who received study treatment and had post-baseline IELT data available based on the dose actually received by the participants. Number analyzed is the number of participants with available data at the given time-point.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | OnabotulinumtoxinA Dose 1 | OnabotulinumtoxinA Dose 2 | OnabotulinumtoxinA Dose 3 | OnabotulinumtoxinA Dose 4 | OnabotulinumtoxinA Dose 5 | OnabotulinumtoxinA Dose 6 | Placebo
Number analyzed (Participants) | 5 | 7 | 8 | 7 | 8 | 7 | 15
seconds
  Baseline: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 15
  Baseline | 37.25 (10.518) | 39.42 (21.504) | 34.41 (10.194) | 38.00 (16.008) | 40.88 (16.435) | 38.75 (15.596) | 37.92 (16.656)
  Change from Baseline to Week 2: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 14
  Change from Baseline to Week 2 | 66.25 (101.132) | 180.31 (317.657) | 24.73 (59.725) | 34.87 (74.842) | 28.04 (31.298) | 55.77 (65.549) | 11.25 (23.985)
  Change from Baseline to Week 4: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 14
  Change from Baseline to Week 4 | 61.94 (100.446) | 176.71 (367.665) | 24.06 (59.472) | 35.00 (73.475) | 28.46 (36.881) | 64.97 (67.471) | 29.30 (69.073)
  Change from Baseline to Week 6: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 14
  Change from Baseline to Week 6 | 61.42 (100.446) | 183.44 (374.404) | 20.75 (55.850) | 36.95 (71.996) | 29.35 (39.334) | 64.49 (66.546) | 47.62 (89.847)
  Change from Baseline to Week 8: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 14
  Change from Baseline to Week 8 | 59.55 (100.896) | 176.59 (349.777) | 17.08 (44.158) | 37.69 (71.873) | 29.48 (44.505) | 65.19 (65.612) | 65.57 (128.470)
  Change from Baseline to Week 10: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 15
  Change from Baseline to Week 10 | 56.13 (101.447) | 170.65 (331.039) | 15.55 (39.149) | 37.45 (71.782) | 27.49 (45.365) | 63.91 (67.725) | 68.26 (146.330)
  Change from Baseline to Week 12: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 15
  Change from Baseline to Week 12 | 53.65 (102.527) | 152.74 (295.219) | 12.95 (30.930) | 28.32 (48.965) | 27.51 (48.720) | 66.01 (71.489) | 68.49 (151.680)
Statistical Analysis 1: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 versus (vs) Placebo at Week 2; Test type: Superiority; p = 0.184, ANCOVA — Least square mean and one-sided p-value of mean difference vs placebo for each active OnabotulinumtoxinA dose level is calculated from the ANCOVA Model with treatment as the fixed effect and baseline average IELT as the covariate; Least square mean difference = 55.33
Statistical Analysis 2: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 2; Test type: Superiority; p = 0.002, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 170.21
Statistical Analysis 3: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 2; Test type: Superiority; p = 0.404, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 12.73
Statistical Analysis 4: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 2; Test type: Superiority; p = 0.328, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 24.23
Statistical Analysis 5: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 2; Test type: Superiority; p = 0.362, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 18.48
Statistical Analysis 6: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 2; Test type: Superiority; p = 0.203, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 45.42
Statistical Analysis 7: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 4; Test type: Superiority; p = 0.322, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 33.05
Statistical Analysis 8: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 4; Test type: Superiority; p = 0.015, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 148.86
Statistical Analysis 9: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 4; Test type: Superiority; p = 0.541, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -6.20
Statistical Analysis 10: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 4; Test type: Superiority; p = 0.459, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 6.47
Statistical Analysis 11: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 4; Test type: Superiority; p = 0.491, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 1.32
Statistical Analysis 12: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 4; Test type: Superiority; p = 0.281, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 36.80
Statistical Analysis 13: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 6; Test type: Superiority; p = 0.424, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 14.12
Statistical Analysis 14: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 6; Test type: Superiority; p = 0.026, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 136.96
Statistical Analysis 15: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 6; Test type: Superiority; p = 0.670, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -27.62
Statistical Analysis 16: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 6; Test type: Superiority; p = 0.561, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -10.06
Statistical Analysis 17: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 6; Test type: Superiority; p = 0.604, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -16.58
Statistical Analysis 18: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 6; Test type: Superiority; p = 0.394, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 17.76
Statistical Analysis 19: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 8; Test type: Superiority; p = 0.532, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -5.94
Statistical Analysis 20: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 8; Test type: Superiority; p = 0.058, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 111.27
Statistical Analysis 21: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 8; Test type: Superiority; p = 0.778, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -48.65
Statistical Analysis 22: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 8; Test type: Superiority; p = 0.662, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -27.74
Statistical Analysis 23: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 8; Test type: Superiority; p = 0.712, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -35.72
Statistical Analysis 24: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 8; Test type: Superiority; p = 0.501, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -0.18
Statistical Analysis 25: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 10; Test type: Superiority; p = 0.565, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -12.14
Statistical Analysis 26: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 10; Test type: Superiority; p = 0.071, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 102.44
Statistical Analysis 27: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 10; Test type: Superiority; p = 0.799, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -52.81
Statistical Analysis 28: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 10; Test type: Superiority; p = 0.681, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -30.81
Statistical Analysis 29: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 10; Test type: Superiority; p = 0.741, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -40.68
Statistical Analysis 30: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 10; Test type: Superiority; p = 0.526, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -4.33
Statistical Analysis 31: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 12; Test type: Superiority; p = 0.584, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -14.76
Statistical Analysis 32: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 12; Test type: Superiority; p = 0.101, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = 84.09
Statistical Analysis 33: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 12; Test type: Superiority; p = 0.823, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -55.14
Statistical Analysis 34: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 12; Test type: Superiority; p = 0.741, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -40.18
Statistical Analysis 35: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 12; Test type: Superiority; p = 0.756, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -41.31
Statistical Analysis 36: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 12; Test type: Superiority; p = 0.517, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least square mean difference = -2.57

3. Secondary Outcome: Change From Baseline in Geometric Mean IELT
Description: IELT, the time from vaginal penetration to ejaculation, was measured by a stopwatch and was recorded in the SID. The Logarithm Value of the Geometric Mean of each individual participant's IELT recorded in the SID up to each time point was calculated. The mean and SD of log-transformed geometric mean IELTs were then calculated for each treatment group. An ANCOVA Model with treatment as the fixed effect and baseline geometric mean IELT as the covariate was used for analyses. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Weeks 2, 4, 6, 8, and 10
Population: The mITT population included all randomized participants who received study treatment and had post-baseline IELT data available based on the dose actually received by the participant. Number analyzed is the number of participants with available data at the given time-point.
Measure: Mean (Standard Deviation); unit: log(seconds)
Arm/Group | OnabotulinumtoxinA Dose 1 | OnabotulinumtoxinA Dose 2 | OnabotulinumtoxinA Dose 3 | OnabotulinumtoxinA Dose 4 | OnabotulinumtoxinA Dose 5 | OnabotulinumtoxinA Dose 6 | Placebo
Number analyzed (Participants) | 5 | 7 | 8 | 7 | 8 | 7 | 15
log(seconds)
  Baseline: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 15
  Baseline | 3.57 (0.283) | 3.50 (0.631) | 3.46 (0.371) | 3.52 (0.531) | 3.53 (0.475) | 3.54 (0.505) | 3.46 (0.610)
  Change from Baseline to Week 2: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 14
  Change from Baseline to Week 2 | 0.76 (1.014) | 0.95 (1.497) | 0.26 (0.677) | 0.34 (0.690) | 0.47 (0.604) | 0.62 (0.623) | 0.19 (0.486)
  Change from Baseline to Week 4: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 14
  Change from Baseline to Week 4 | 0.70 (1.000) | 0.77 (1.505) | 0.18 (0.879) | 0.33 (0.616) | 0.38 (0.481) | 0.61 (0.618) | 0.22 (0.627)
  Change from Baseline to Week 6: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 14
  Change from Baseline to Week 6 | 0.70 (0.999) | 0.83 (1.513) | 0.08 (0.971) | 0.36 (0.629) | 0.36 (0.483) | 0.59 (0.722) | 0.36 (0.524)
  Change from Baseline to Week 8: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 14
  Change from Baseline to Week 8 | 0.67 (1.007) | 0.79 (1.525) | 0.05 (0.968) | 0.37 (0.627) | 0.36 (0.522) | 0.61 (0.682) | 0.44 (0.567)
  Change from Baseline to Week 10: number analyzed (Participants) | 5 | 6 | 8 | 7 | 8 | 7 | 15
  Change from Baseline to Week 10 | 0.60 (1.009) | 0.80 (1.503) | 0.07 (0.905) | 0.37 (0.624) | 0.32 (0.512) | 0.56 (0.727) | 0.44 (0.603)
Statistical Analysis 1: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 2; Test type: Superiority; p = 0.079, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.59
Statistical Analysis 2: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 2; Test type: Superiority; p = 0.025, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.77
Statistical Analysis 3: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 2; Test type: Superiority; p = 0.417, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.07
Statistical Analysis 4: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 2; Test type: Superiority; p = 0.330, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.16
Statistical Analysis 5: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 2; Test type: Superiority; p = 0.199, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.30
Statistical Analysis 6: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 2; Test type: Superiority; p = 0.113, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.45
Statistical Analysis 7: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 4; Test type: Superiority; p = 0.127, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.50
Statistical Analysis 8: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 4; Test type: Superiority; p = 0.087, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.56
Statistical Analysis 9: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 4; Test type: Superiority; p = 0.543, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.04
Statistical Analysis 10: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 4; Test type: Superiority; p = 0.377, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.12
Statistical Analysis 11: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 4; Test type: Superiority; p = 0.321, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.17
Statistical Analysis 12: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 4; Test type: Superiority; p = 0.149, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.40
Statistical Analysis 13: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 6; Test type: Superiority; p = 0.215, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.35
Statistical Analysis 14: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 6; Test type: Superiority; p = 0.126, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.47
Statistical Analysis 15: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 6; Test type: Superiority; p = 0.774, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.28
Statistical Analysis 16: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 6; Test type: Superiority; p = 0.495, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.01
Statistical Analysis 17: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 6; Test type: Superiority; p = 0.495, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.00
Statistical Analysis 18: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 6; Test type: Superiority; p = 0.274, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.23
Statistical Analysis 19: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 8; Test type: Superiority; p = 0.308, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.22
Statistical Analysis 20: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 8; Test type: Superiority; p = 0.205, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.34
Statistical Analysis 21: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 8; Test type: Superiority; p = 0.849, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.39
Statistical Analysis 22: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 8; Test type: Superiority; p = 0.571, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.07
Statistical Analysis 23: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 8; Test type: Superiority; p = 0.592, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.09
Statistical Analysis 24: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 8; Test type: Superiority; p = 0.340, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.16
Statistical Analysis 25: Comparison: OnabotulinumtoxinA Dose 1 vs Placebo; OnabotulinumtoxinA Dose 1 vs Placebo at Week 10; Test type: Superiority; p = 0.360, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.16
Statistical Analysis 26: Comparison: OnabotulinumtoxinA Dose 2 vs Placebo; OnabotulinumtoxinA Dose 2 vs Placebo at Week 10; Test type: Superiority; p = 0.192, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.35
Statistical Analysis 27: Comparison: OnabotulinumtoxinA Dose 3 vs Placebo; OnabotulinumtoxinA Dose 3 vs Placebo at Week 10; Test type: Superiority; p = 0.843, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.37
Statistical Analysis 28: Comparison: OnabotulinumtoxinA Dose 4 vs Placebo; OnabotulinumtoxinA Dose 4 vs Placebo at Week 10; Test type: Superiority; p = 0.572, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.07
Statistical Analysis 29: Comparison: OnabotulinumtoxinA Dose 5 vs Placebo; OnabotulinumtoxinA Dose 5 vs Placebo at Week 10; Test type: Superiority; p = 0.628, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = -0.12
Statistical Analysis 30: Comparison: OnabotulinumtoxinA Dose 6 vs Placebo; OnabotulinumtoxinA Dose 6 vs Placebo at Week 10; Test type: Superiority; p = 0.380, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least square mean difference = 0.12

ADVERSE EVENTS:
Time Frame: First dose and for at least 28 days after the last dose of study medication (Up to 26 Weeks in the Randomized-treatment Period and Up to 17 Weeks in the Open-Label Period)
Description: A treatment-emergent adverse event (TEAE) was an adverse event with onset on or after the initiation of study treatment or an adverse event with onset prior to study treatment that worsened in severity or became serious after the initiation of study treatment.
  Safety Population included all treated participants.
Groups:
- OnabotulinumtoxinA Dose 2: OnabotulinumtoxinA Dose 2 injected into specified muscle per protocol on Day 1.
Arm/Group | OnabotulinumtoxinA Dose 1 | OnabotulinumtoxinA Dose 2 | OnabotulinumtoxinA Dose 3 | OnabotulinumtoxinA Dose 4 | OnabotulinumtoxinA Dose 5 | OnabotulinumtoxinA Dose 6 | Placebo | OnabotulinumtoxinA Dose 2 (Open-label Period)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7 | 0/8 | 0/8 | 0/8 | 0/8 | 0/15 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/8 | 0/8 | 0/8 | 0/8 | 0/15 | 0/8
Other Adverse Events (participants affected / at risk) | 3/5 | 2/7 | 1/8 | 2/8 | 3/8 | 4/8 | 12/15 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA Dose 1 (N=5) | OnabotulinumtoxinA Dose 2 (N=7) | OnabotulinumtoxinA Dose 3 (N=8) | OnabotulinumtoxinA Dose 4 (N=8) | OnabotulinumtoxinA Dose 5 (N=8) | OnabotulinumtoxinA Dose 6 (N=8) | Placebo (N=15) | OnabotulinumtoxinA Dose 2 (Open-label Period) (N=8)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Penis injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Semen volume decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enuresis (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychogenic erectile dysfunction (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Terminal dribbling (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Epididymal tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ejaculation failure (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT01917006/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT01917006/SAP_001.pdf